CLINICAL TRIAL: NCT04234243
Title: HIPEC in Ovarian Cancer: The First Case Control Study in Mexican Patients With 10-year Follow-up
Brief Title: HIPEC in Ovarian Cancer, Case-Controls Study With 10-years Follow up
Status: Completed | Type: Observational
Sponsor: Instituto de Seguridad Social del Estado de Mexico y Municipios (Other Government)
Responsible Party: Principal Investigator, Juan Manuel Medina Castro, Peritoneal Malignacy neoplasm coordinator, Instituto de Seguridad Social del Estado de Mexico y Municipios
Other Study IDs: COE-UEI/05/PT/2016
Record Dates: First submitted 2020-01-10; First posted 2020-01-21 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Ovarian Cancer; HIPEC
Keywords: HIPEC
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIPEC: women, with ovarian cancer stage III-IV or recurrent with carcinomatosis treated with cytoreduction and HIPEC
  Interventions: Procedure: cytoreduction and HIPEC
- No HIPEC: women, with ovarian cancer stage III-IV or recurrent with carcinomatosis, treated with systemic chemotherapy only

INTERVENTIONS:
Procedure: cytoreduction and HIPEC — cytoreduction CCR 0-1, and HIPEC close technique
  Groups: HIPEC

SUMMARY:
Objectives:

Compare overall survival (OS) and progression-free survival (PFS) among ovarian cancer patients who underwent into cytoreduction and HIPEC procedure vs patients who only received systemic chemotherapy in a 10-years follow up of a case-control study

Methods:

Cases were defined as patients treated by cytoreduction and HIPEC, and were matched (1:2) with patients treated with chemotherapy only, defined as controls. PFS and OS in the two groups were measured and compared. PFS was calculated from initiation of treatment to progression, death or to the last known follow-up. OS was calculated from initiation of treatment to death or to the last known follow-up.

DETAILED DESCRIPTION:
Epithelial ovarian cancer has the highest mortality of all gynecologic tumors in the world wide. Patients are diagnosed with International Federation of Gynecology and Obstetrics (FIGO) stage III to IV disease in 75%. The 10-year survival of women with advanced-stage ovarian cancer is 10% to 15% and has not improve in the past 20 years. Despite treatment with maximal cytoreductive surgery (CRS) and platinum-based chemotherapy, approximately 70% of patients with advanced-stage disease relapse within 18 months. Given this high number of recurrences, new approaches are needed to improve outcomes for these patients. Historically, peritoneal carcinomatosis represents a devastating form of cancer progression with a very poor prognosis.

Objectives:

Compare overall survival (OS) and progression-free survival (PFS) among ovarian cancer patients who underwent into cytoreduction and HIPEC procedure vs patients who only received systemic chemotherapy in a 10-years follow up of a case-control study

Methods:

Cases were defined as patients treated by cytoreduction and HIPEC, and were matched (1:2) with patients treated with chemotherapy only, defined as controls. PFS and OS in the two groups were measured and compared. PFS was calculated from initiation of treatment to progression, death or to the last known follow-up. OS was calculated from initiation of treatment to death or to the last known follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Epithelial ovarian cancer confirmed
* FIGO stage III-IV or carcinomatosis recurrence
* No comorbidities or controlled comorbidities
* ECOG 0-2

Exclusion Criteria:

* without carcinomatosis

Ages: 18 Years to 72 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIPEC population: 46 patients No HIPEC population : 92 patients
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
free overall survival | 10 years
  survillance from HIPEC procedure/IV chemotherapy for carcinomatosis, to death date or last consultation (months) Kaplan Meier curve
free recurrence survival | 10 years
  survillance from HIPEC procedure/IV chemotherapy for carcinomatosis, to recurrence date (months) Kaplan Meier curve

SECONDARY OUTCOMES:
factors associated with survival | 10 years
  histological and clinical factors associated with survival. uni and multivariate analysis (X2, Cox, U Mann-Witney)